CLINICAL TRIAL: NCT04520711
Title: Hotspot TCR-T: A Phase I/Ib Study of Adoptively Transferred T-cell Receptor Gene-engineered T Cells (TCR-T) Targeting Tumor-Specific Neoantigens, With in Vivo CD40 Activation and PD-1 Blockade, for Patients With Incurable Cancers (2020000584)
Brief Title: Hotspot TCR-T: A Phase I/Ib Study of Adoptively Transferred T-cell Receptor Gene-engineered T Cells (TCR-T)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020000584
Record Dates: First submitted 2020-08-15; First posted 2020-08-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Malignant Epithelial Neoplasms
MeSH Terms: conditions — Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CDX-1140 + TCR-T + Pembro (Experimental): Patients will receive CDX-1440, TCR-T, and pembrolizumab.
  Interventions: Biological: TCR-transduced T cells; Drug: CDX-1140; Drug: Pembrolizumab

INTERVENTIONS:
Biological: TCR-transduced T cells — TSA-reactive TCR-engineered T cells
Drug: CDX-1140 — Recombinant fully human IgG2κ monoclonal antibody
Drug: Pembrolizumab — Humanized immunoglobulin G4 (IgG4) monoclonal antibody

SUMMARY:
This is a phase I/Ib study of adoptively transferred T-cell receptor gene-engineered T cells (TCR-T) targeting tumor-specific antigens, with in vivo CD40 activation and PD-1 blockade, for patients with incurable cancers. The study design is a safety lead-in TCR-T with CD40/PD-1 (3+3), followed by Simon's Two-Stage expansion design, 80% power and 5% one-sided alpha: stage-one futility assessment at n = 10; stage-two assessment at n = 22, (accrual up to 24 to allow for potential study drop-out).

DETAILED DESCRIPTION:
Patients will be infused with T cells engineered to express TCRs targeting one to five tumor-specific antigens expressed by their autologous tumor. The number of T cells infused will range from 1e9 to 1e11. Monoclonal antibodies targeting PD-1 (pembrolizumab) and CD40 (CDX-1140, Celldex Therapeutics)43 will be administered, in that order, starting within 24 hours of cell infusion and re-administered at approximately 3 week intervals. Clinic visits will include longitudinal evaluation of toxicities and monitoring of immunological parameters. The presence or absence of replication competent retrovirus (RCR) will be evaluated for the first year following adoptive cell transfer, or longer, if there is evidence of RCR.

Tumor Response assessment by RECIST 1.1 is performed every 9-12 weeks. Study treatment continues until progression. Option repeat TCR-T infusion is allowed and in addition may incorporate preconditioning chemotherapy using a de-intensified non-myeloablative (NMA) regimen consisting of a single dose of gemcitabine and a single dose of either cyclophosphamide or epirubicin, designed to elicit immunogenic cell death and transient lymphopenia.

The primary objective of this study is to determine the safety of the adoptive transfer of TCR-gene engineered T cells targeting TSA in combination with CD40 and PD-1 immunotherapy. The secondary objective is to determine whether this therapy can mediate objective clinical responses as determined by objective criteria (e.g. RECIST 1.1). The study will also characterize the differentiation and functional state of the TCR-gene modified T cells before and after cell therapy and monitor their persistence in the patient after treatment. Up to 24 patients will be enrolled in this study. Based on published trials treating patients with TCR-transduced T cells, adverse events such as fever, chills, dyspnea, hypotension, fatigue, edema, rash, and rarely acute cytokine release syndrome, may occur.

Clinical and immunological data will be analyzed which will determine whether this therapy is safe and effective, and whether there are biomarkers or immunological signatures that correlate to efficacy and/or lack of efficacy. This data will determine whether additional studies are warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and older with metastatic or locoregionally advanced epithelial cancers, that are considered incurable.
2. Confirmation by Tran Laboratory of neoantigen-reactive TCR(s) suitable for TCR-gene therapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
4. Laboratory values:

   * WBC ≥ 2000/uL
   * Neutrophils ≥ 1000/uL
   * Hgb > 8.0 g/dl (patients may be transfused to reach this level)
   * Platelets > 100,000 cells/mm3
   * Creatinine ≤ 2.0 mg/dL
   * AST & ALT ≤ 2.5 × ULN
   * Alkaline phosphatase ≤ 2.5 × ULN
   * Total bilirubin ≤ 2 × ULN (except patients with Gilbert's syndrome, who must have a total bilirubin ≤ 3.0 mg/dL). If total bilirubin is >1.5, conjugated bilirubin must be ≤ ULN (conjugated bilirubin only needs to be tested if total bilirubin exceeds ULN). If there is no institutional ULN, then conjugated bilirubin must be < 40% of total bilirubin.
5. Patients positive for hepatitis B core antibody (anti-HBc, total), are eligible only if HBV DNA is non- detectable by qPCR.
6. Patients positive for hepatitis C virus (HCV) antibody are eligible only if HCV RNA is non-detectable by qPCR.
7. Patients known positive for HIV 1/2 antibodies, are eligible if ARV treatment compliant with documented stable absolute CD4 count > 300 cells/mm3 for at least 6 months and undetectable viral load.
8. Women of childbearing potential must have negative serum bHCG pregnancy test ≤ 24 hours prior to start of study treatment.
9. Ability to give informed consent and comply with the protocol.
10. Anticipated lifespan greater than 12 weeks.
11. Men and women of childbearing potential must agree to take appropriate pregnancy precautions during treatment and through 180 days after last dose of study treatment. Patients and/or partners who are surgically sterile or postmenopausal (defined by 12 or more consecutive months with no menstruation, or surgically sterile) are exempt from this requirement. Males must agree not to donate sperm for at least 90 days after discontinuing study treatment.

Exclusion Criteria:

1. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
2. Receipt of any investigational anticancer therapy during the last 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study treatment. Receipt of any prior anti-CD40 therapy.
3. Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment, within 21 days (6 weeks for nitrosoureas) or at least 5 half-lives (whichever is longer) prior to the first dose of study treatment. Concurrent use of 4. hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

5. Local treatment of isolated lesions for palliative intent is acceptable (e.g., local surgery or radiotherapy), excluding target lesions, Palliative radiation therapy cannot be administered less than 1 week prior to the first dose of study treatment.

6. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug. Participants must have recovered (to a grade 1 or lower) from all radiation-related toxicities, not require corticosteroids for this purpose and not have had radiation pneumonitis.

7. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study treatment. Note: Local surgery of isolated lesions for palliative intent is acceptable.

8. History of organ transplant, including allogeneic stem cell transplantation. 9. History of (non-infectious) pneumonitis/interstitial lung disease or current pneumonitis/interstitial lung disease, including grade 1 pneumonitis (asymptomatic; clinical or diagnostic observation only; intervention not indicated).

10. Uncontrolled intercurrent illness as deemed by the investigator, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, unstable cardiac arrhythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.

11. History of another primary malignancy except for:

* Malignancy treated with curative intent and with no known active disease ≥1 year before the first dose of investigational product and of low potential risk for recurrence.
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease (per investigator discretion).
* Adequately treated carcinoma in situ without evidence of disease (per investigator discretion) 12. History of leptomeningeal carcinomatosis 13. Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients whose brain metastases have been treated may participate provided they show radiographic stability (imaging at least four weeks apart showing no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤ 10mg/day of prednisone or its equivalent and anti-seizure medications for at least 14 days prior to the start of treatment. Patients on a stable dose of seizure medicines for epilepsy unrelated to cancer are eligible for the trial.

  14. History of active primary immunodeficiency. 15. Active tuberculosis infection (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice).

  16. Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg/day of prednisone or equivalent).:
* Autoimmune disease that is not active (in remission), but in the judgment of the investigator could risk substantial morbidity in the event of relapse, may be grounds for exclusion. This can include a prior history of pneumonitis or other autoimmune sequelae of prior immunotherapy.
* Physiologic corticosteroid replacement therapy at doses > 10 mg/day of prednisone or equivalent for adrenal or pituitary insufficiency and in the absence of active autoimmune disease is permitted.
* Participants with asthma that requires intermittent use of bronchodilators, inhaled steroids, or local steroid injections may participate.
* Participants using topical, ocular, intra-articular, or intranasal steroids (with minimal systemic absorption, per investigator discretion) may participate.

  17. Brief courses of corticosteroids for prophylaxis (e.g., contrast dye allergy) or study treatment-related standard premedication are permitted.

  18. Receipt of live attenuated vaccine within 28 days prior to the first dose of study treatment. Note: patients should not receive live vaccine during study treatment and up to 30 days after the last dose of study treatment.

  19. Known allergy or hypersensitivity to study drug(s) or compounds of similar biologic composition to the study drug(s), or any of the study drug excipients.

  20. Any unresolved NCI CTCAE Grade ≥2 toxicities from prior anti-cancer therapy (see above for radiotherapy consideration) with the exception of vitiligo or alopecia, and per investigator discretion for laboratory values not defined in the inclusion criteria.

  21. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Principal Investigator or one of the Co-Principal Investigators.

  22. Patients with irreversible toxicity not reasonably expected to be exacerbated by study treatment may be included only after consultation with the Principal Investigator or one of the Co-Principal Investigators.

  23. Immune-related toxicity during prior checkpoint inhibitor therapy for which permanent discontinuation of therapy is recommended (per product label or consensus guidelines) OR any immune-related toxicity requiring intensive or prolonged immunosuppression to manage (with the exception of endocrinopathy that is well controlled on replacement hormones).

  24. Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension or arrhythmia, congestive heart failure (NYHA Class III or IV) related to primary cardiac disease, uncontrolled ischemic or severe valvular heart disease. Patients with a history of myocardial infarction, cerebral vascular accident, thrombosis or pulmonary embolus within 12 months prior to the first dose of study treatment are excluded from this study.

  25. Any other acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial.

  26. Women who are pregnant, lactating or expecting to conceive, or men who father children within the projected duration of the study.

  27. Unable or unwilling to comply with study requirements, including follow-up visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety, tolerability and DLTs of combinatorial adoptively transferred T-cell receptor gene-engineered T cells (TCR-T) with in vivo CD40 activation and PD-1 blockade, for patients with incurable cancers | 2 years
  Analysis of adverse events

SECONDARY OUTCOMES:
Objective response rate | 2 years
  percentage of subjects having CR or PR
Duration of response | 2 years
  the time from the earliest date of disease response (CR or PR) until earliest date of disease progression or death due to any cause
Clinical benefit rate | 2 years
  percentage of subjects having CR, PR, or SD (with minimum duration > 4 months)
Overall survival | 2 years
  determined by survival follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rom Leidner, MD, Principal Investigator — Providence Health & Services; Eric Tran, PhD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No